CLINICAL TRIAL: NCT03265379
Title: Improving Quality of Life for Patients With Breast Cancer Invading the Chest Wall: A Prospective Registry For Patients Undergoing Full Thickness Chest Wall Resection
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-5560
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients with an isolated recurrence in the chest wall
  Interventions: Other: FACT-B and Brief Pain Inventory
- distant metastatic disease is present but who undergo FTCWR
  Interventions: Other: FACT-B and Brief Pain Inventory
- patient with primary tumor, no distant ds, failed conventional
  Interventions: Other: FACT-B and Brief Pain Inventory
- patients refusing to undergo surgery
  Interventions: Other: FACT-B and Brief Pain Inventory

INTERVENTIONS:
Other: FACT-B and Brief Pain Inventory — Quality of Life Questionnaires

SUMMARY:
Although chest wall recurrence of breast cancer is uncommon, it represents a difficult clinical scenario. The role of full thickness chest wall resection (FTCWR) for breast cancer recurrence in the chest wall is controversial and is complicated by the fact that no prospective evidence exists evaluating the utility of FTCWR in prolonging survival or improving health related quality of life (HRQOL) and thus, there is a lack of evidence to guide treatment decisions. Gathering HRQOL, local-regional recurrence (LRR) and survival data in a prospective fashion is thus critical in this population. Therefore, we designed a prospective trial to evaluate the outcomes for FTCWR in terms of LRC and HRQOL, and short-term morbidity and mortality, with secondary focus on potential long-term overall survival benefit.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized cohort study for patients with chest wall-recurrent/invasive breast cancer treated with full thickness chest wall resection (FTCWR), chemotherapy and/or radiation. The design of this study was created using the framework for surgical trials set out by the IDEAL collaboration (Idea, Development, Exploration, Assessment, Long-Term follow up), 14 after a systematic evaluation of the current literature had been completed. Given that no prospective evidence exists in this patient population and based on the IDEAL framework, this study is designed to create a prospective registry.

Data on the efficacy of the standard interventions (surgery, chemotherapy, radiation) will be evaluated using 'global criteria', that is, the data that will be collected via the scores on the FACT-B, the Brief Pain Inventory, and the specific cancer outcomes as outlined previously (local regional recurrence (LRC), overall survival, short term morbidity and mortality as well as disease-free survival).

The primary objective is to measure the differences in Functional Assessment of Cancer Therapy - Breast (FACT-B) scale scores from baseline to 6 month evaluation.

In addition to measuring health related quality of life (HRQOL) at 6 months, differences in the FACT-B scale at 1-month, 3-months and 1-year postoperatively will be examined. Rates of LRC, defined as local recurrence in the ipsilateral chest wall, axilla, infra- or supraclavicular region at 1, 2, 3 and 5-years postoperatively will be measured, as well as thirty and ninety-day morbidity and mortality (to be classified using the Thoracic Morbidity and Mortality (TM and M) classification system). As well, data will be collected on overall survival, measured as the proportion of patients surviving to at 1-year, 2-years, 3-years and 5 years postoperatively. Lastly, data will be collected on disease-free survival, defined as any evidence of systemic recurrence plus LRR at 1-year, 2-years, 3-years and 5-years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Breast cancer with invasion of the chest wall (ribs, para-costal soft tissue, intercostal muscle or soft-tissue) that is:

   1. Radiologically proven on cross-sectional imaging
   2. Histologically proven
3. Medically fit for surgery
4. >1 year disease-free interval (between initial treatment and recurrence) for patients with local recurrence

Exclusion Criteria:

1. Medically inoperable due to co-morbidity or other contraindication to surgery
2. Technically unresectable disease
3. Ineligible for chemotherapy
4. ECOG performance status >2
5. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest wall-recurrent/invasive breast cancer treated with FTCWR, chemotherapy and/or radiation.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2030-08-22 (Estimated); Study Completion 2030-08-22 (Estimated)

PRIMARY OUTCOMES:
differences in Functional Assessment of Cancer Therapy - Breast (FACT-B) scale scores | from baseline to 6 month evaluation

SECONDARY OUTCOMES:
FACT-B scale | 1-month, 3-months and 1-year postoperatively
Local Recurrence | 1, 2, 3 and 5-years postoperatively
Morbidity and mortality | 90 days post op
Overall Survival | 1-year, 2-years, 3-years and 5 years postoperatively
Disease Free Survival | 1-year, 2-years, 3-years and 5 years postoperatively
Brief Pain Inventory | 1 month, 3 months, 6 months and 1 year postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Shaf Keshavjee, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network (Toronto General Hospital and Princess Margaret Cancer Centre), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No